CLINICAL TRIAL: NCT06179212
Title: Comparing VO2 Peak Values of Exercise Testing Protocols for Females and Males With CAD
Brief Title: Exercise Testing Protocols for Females and Males With CAD
Acronym: PACED
Status: Not yet recruiting | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 20230327-01H
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CPETs: Patients will perform all 4 maximal cardiopulmonary exercise tests in randomized order. The protocols they will perform are: Modified Bruce, modified Naughton, modified Balke and the UOHI Slow Ramp.
  Interventions: Diagnostic Test: Exercise Tests

INTERVENTIONS:
Diagnostic Test: Exercise Tests — Patients will complete 4 different cardiopulmonary exercise tests in random order.

SUMMARY:
The aim of this study is to determine if the test that allows males to achieve a higher VO2 (a measure of oxygen use during exercise) is different for females. The purpose of this study is to test 4 different exercise testing protocols to compare measured oxygen consumption in females and males with CAD (disease caused by the buildup of plaque in the artery walls which can lead to insufficient amounts of blood, nutrients and oxygen being supplied to the heart). The 4 exercise tests that will be completed on the treadmill are the modified Balke, modified Bruce, modified Naughton and University of Ottawa Heart Institute Slow Ramp protocols. Each test has a different stage duration (the amount of time that the test remains at a pre-determined speed and incline), and incremental increase in speed and incline.

The main purpose of this study is to compare VO2 peak (the maximal amount of oxygen utilized during the exercise test) of females and males with CAD in 4 different exercise protocols. For example, the investigators will find out:

1. which exercise protocol is more likely to achieve a higher peak V̇O2 in females and which protocol is more likely to achieve a higher peak V̇O2 in males,
2. if enjoyment affects the duration of the test, and
3. how different exercise test protocols will provide different results of maximal oxygen used by the participant's body during the exercise test.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older;
2. previous CAD diagnosis by a physician;
3. can perform a CPET until volitional exhaustion;
4. are able to self-ambulate on a treadmill;
5. are at least 8 weeks post cardiovascular event or procedure (i.e., percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG)); and,
6. are able to provide written informed consent.

Exclusion Criteria:

1. cannot speak, read, write, or understand English or French;
2. currently not enrolled in a CR program;
3. have recently changed (or planning to change) PA levels within the previous 4 weeks (as this may impact the ability to compare outcomes between exercise testing protocols);
4. have heart failure with an ejection fraction <45% (indication of possible cardiomyopathy);6
5. have an arrythmia (relative contraindication for exercise testing),6 peripheral artery disease, valvular disease, severe aortic stenosis, cardiomyopathy, SCAD and/or COPD (contraindications for maximal exercise testing);
6. has an ICD;
7. is pregnant (sustained vigorous exercise in pregnant women may induce fetal bradycardia)
8. is unable to complete submaximal exercise testing (i.e., treadmill, due to musculoskeletal limitations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults older than 18 years of age and have been diagnosed with CAD.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-05-21 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Oxygen Consumption (VO2) | Week 1 to week 4 (measured weekly, at every appointment)
  V̇O2 will be measured continuously throughout the treadmill CPET. Peak V̇O2, defined as the highest V̇O2 value that is achieved over a 20-s period during the last minute of the CPET. V̇O2 will be measured throughout each test by a metabolic system (Parvo Medics TrueOne 2400).

SECONDARY OUTCOMES:
Cardiometabolic health indicators - Blood pressure (BP) | Week 1 to week 4 (measured weekly, at every appointment)
  Resting BP (mmHg) will be measured from a seated position using an automated BP monitor. BP will be measured manually using a BP cuff every 2 stages throughout the CPET using an automated BP monitor. Recovery BP will be measured after the completion of the test from a seated position using the automated BP monitor.
Cardiometabolic health indicators - Heart Rate (HR) | Week 1 to week 4 (measured weekly, at every appointment)
  Heart rate will be measured from a seated position using an automated BP monitor. HR will be measured continuously throughout the CPET using a 4-lead electrocardiogram connected to a metabolic system. Recovery HR will be measured after the completion of the test from a seated position using the automated BP monitor.
Cardiometabolic health indicators - Body mass index | Week 1 to week 4 (measured weekly, at every appointment)
  Height (cm) and body mass (kg) will be measured to compute body mass index (kg/m2).
Cardiometabolic health indicators - Fat mass | Week 1 to week 4 (measured weekly, at every appointment)
  Fat mass (kg) and fat-free mass (kg) will be measured using bioelectrical impedance.
Cardiometabolic health indicators - Waist circumference | Week 1 to week 4 (measured weekly, at every appointment)
  Waist circumference will be measured using standardized procedures (2 repeated measures using a tape; in centimeters).
Cardiometabolic health indicators - Height | Week 1 to week 4 (measured weekly, at every appointment)
  Height will be measured using standardized procedures (2 repeated measures using a tape; in centimeters).
Blood Lactate | Week 1 to week 4 (measured weekly, at every appointment)
  Blood lactate (mmol/L) will be measured in the last 30s of every test stage throughout the test using a blood lactate analyzer.
Rating of perceived exertion (RPE) | Week 1 to week 4 (measured weekly, at every appointment)
  Measured at the end of every stage using the validated Borg 6-20 rating of perceived exertion scale. This scale measures how physically exerted an individual feels. 6 is complete rest (i.e., no exertion, ex: sitting in a chair not moving and relaxed), 20 is perceived maximal exertion of effort. These values are perceived measures of effort and will increase as the exercise test progresses and gets harder for the patient.
Test duration | Week 1 to week 4 (measured weekly, at every appointment)
  Measured using portable metabolic system that is connected to a computer. The duration of the test will be recorded.
Reason for test termination | Week 1 to week 4 (collected weekly, at every appointment)
  Reason for test termination will be collected subjectively by asking the patient (i.e., fatigue, muscular limitation, etc.)
Physical activity enjoyment | Week 1 to week 4 (collected weekly, at every appointment)
  This is a subjective questionnaire that measures the extent to which the patient enjoyed participating in the test.
Most enjoyed test | Week 4 - collected at the patient's last appointment
  Using a feedback questionnaire, the test that was most frequently ranked the most enjoyed by patients will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation